CLINICAL TRIAL: NCT05872971
Title: Dry Needling vs Lasertherapy in Greater Trochanteric Pain Syndrome (GTPS): Randomized Clinical Trial
Brief Title: Dry Needling and Lateral Hip Pain (GTPS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, advisor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dry Needling e quadril
Record Dates: First submitted 2023-04-25; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Trochanteric Bursitis
Keywords: lateral hip pain; trochanteric bursitis; greater trochanteric gluteal syndrome
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: This is a randomized blind clinical trial, with a longitudinal characteristic in the area of physiotherapy and orthopedics. The intervention will consist of 6 weeks, 2 times a week, and the variables of interest will be measured in the pre-treatment period, after the first week, after the third week of treatment, after the end of treatment and after that, there will be a follow up of eight and twelve weeks after treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluations of the participants and the analysis of the data will be carried out by a researcher blind to the allocation of the subjects in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): The technique will be used by a physiotherapist experienced in orthopedic conditions and with specific training in DN.
  Interventions: Device: Dry Needling
- Lasertherapy (Active Comparator): The application of the Laser will be performed by a physiotherapist specialized in traumato-orthopedics.
  Interventions: Device: Lasertherapy

INTERVENTIONS:
Device: Dry Needling — Dry Needling: The technique will be used by a physiotherapist experienced in orthopedic conditions and with specific training in DN. The application will be through the deep technique, above 10mm deep, the therapist will score trigger points regions of the muscles of the posterolateral region of the hip with application duration of 30 to 60 seconds. Eight points of application will be standardized in the region of the muscles of the posterolateral region of the hip.
  Arms: Dry Needling
Device: Lasertherapy — Lasertherapy: The application of the Laser will be performed by a physiotherapist specialized in traumato-orthopedics. The equipment will be infrared laser (904 nm), by point technique. Eight points of application will be standardized in the region of muscles of the posterolateral region of the hip. The time, dose and amounts of application points will be guided according to the dosimetry criteria of the World Association for Photobiomodulation Therapy.
  Arms: Lasertherapy

SUMMARY:
Introduction: Greater Trochanter Pain Syndrome (GTPS) includes a number of disorders involving the lateral hip region, including bursitis, gluteal lacerations, and trigger points in the contractile tissue crossing the hip. As an alternative resource for pain relief, dry needling, known as Dry Needling (DN) is a technique that has been shown to be effective in the treatment of soft tissue injuries and neuromyofascial pain, with positive effects on musculoskeletal conditions. Objective: to compare the administration of ND and laser therapy on the effectiveness of reducing lateral hip pain and improving function in women with GTPS. Materials and methods: The sample will consist of 30 women, aged between 35 and 60, randomized into 2 groups: GND group (n=15) and GLT group (n=15). Participants will complete the sample characterization questionnaire, the numerical pain scale and the VISA Tendinopathy Questionnaire for Greater Trochanteric Pain Syndrome (VISA-G). Subsequently, they will be submitted to evaluation through functional tests sit and stand 30 seconds, Timed up and go test. After the evaluation, they will be submitted to the treatment. The GDN will receive treatment using the technique by a physiotherapist with specific training in NP. The application will be through the deep technique, in the regions of trigger points of muscles of the posterolateral region of the hip with duration of application from 30 to 60 seconds per point, 8 points of application will be standardized, in the region of muscles of the posterolateral region. hip side. The GLT will receive the Laser application by a physiotherapist specialized in traumato-orthopedics. The equipment will be the Infrared Laser (wavelength 904 nm), by punctual technique. Eight application points will be standardized in the muscles region of the posterolateral region of the hip.

DETAILED DESCRIPTION:
If a patient is using an anti-inflammatory, guided by the orthopedist, or a physiotherapy treatment protocol, start only 10 days after the end of the same. As participants, they will be instructed to avoid activities that cause pain during the research period. All others selected until the final evaluation will be discouraged. For all groups, the use of analytical medication prescribed by the orthopedist will be allowed, when requested. As the participants will be asked each session about the use of their analog, the data and the dosage that will occur during the study period will be noted. If necessary, how researchers will contact the orthopedist for information and guidance. If a participant needs to use anti-inflammatory medication during a survey, they will be excluded. The analyzes will be carried out by a blind researcher regarding the allocation of the subjects in each group. Participants who have missing data and those who do not attend all treatment sessions will be included in the analysis.

To establish the results, the following variables will be considered:

* Pain intensity: VAS
* Quality of life: VISA-G questionnaire
* Functional assessment: Soon after, the following functional tests will be performed: 30-second Sit to Stand Test (SL30) and the Timed Up and Go Test (TUG).

The Shapiro-Wilk test will be applied to determine the normality of the sample. Student's t test will be used to compare age, weight, height, body mass index (BMI), and the presence of pain when lying on the hip between groups. The two-way ANOVA test (with Bonferroni post-test) will be used to compare the intra-group and intergroup results, if the data are normal, and will be described as mean and standard deviation. Cohen's D test will be performed to calculate the effect size. Linear correlation between variables will be investigated by Pearson's (or Spearman's) correlation test. If there is a linear correlation between any of the potentially confounding variables, analysis of covariance will be performed using the ANCOVA test. Other necessary analyzes may still be included. The level of statistical significance will be set at p ≤ 0.

ELIGIBILITY:
Inclusion Criteria:

* Lateral hip pain (VAS 3) for at least 3 months
* referring pain to palpation of the insertion of the tendon of the middle and maximum gluteus in the major trochanter
* reproduction of symptoms in at least one of the following tests: 1 - FABER test (Flexion, abduction and external hip rotation) ; 2- Resistive External Rotation Test, 3 - Resistive Isometric Abduction Test , 4 - Unipodal Support Test for 30 seconds.

Exclusion Criteria:

* surgery on lower limbs or spine in the last 12 months

  * symptoms of osteoarthritis or intra-articular disease of the hip (joint block, limited range of motion and difficulty handling socks and clothes)
  * infiltration of the hip with corticosteroids in the last 6 months
  * have received physical therapy for this condition in the past three months
  * participants who need to use anti-inflammatory drugs

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | evaluation before treatment, immediately at the end of treatment and 12 weeks post treatment
  the intensity of your pain using the Visual Analog Pain Scale (VAS), which scores your current pain with scores between 0 and 10. Zero is no pain and 10 is considered unbearable pain

SECONDARY OUTCOMES:
change in hip function | evaluation before treatment, immediately at the end of treatment and after 12 weeks post treatment
  at each assessment, participants will respond to the VISA tendinopathy questionnaire for greater trochanteric pain syndrome, the VISA-G. It consists of eight questions that assess current symptoms with total scores ranging from 0 to 100, with higher scores indicating less pain and better function.
change in lower limb function | evaluation before treatment, immediately at the end of treatment and 12 weeks post treatment
  In each assessment, participants will perform the Timed Up And Go Test (TUG)
change in lower limb function | evaluation before treatment, immediately at the end of treatment and 12 weeks post treatment
  In each assessment, participants will perform the 30'' Sit To Stand Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Christiane Macedo, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Shbeeb MI, Matteson EL. Trochanteric bursitis (greater trochanter pain syndrome). Mayo Clin Proc. 1996 Jun;71(6):565-9. doi: 10.4065/71.6.565. PMID 8642885
- [Background] Del Buono A, Papalia R, Khanduja V, Denaro V, Maffulli N. Management of the greater trochanteric pain syndrome: a systematic review. Br Med Bull. 2012 Jun;102:115-31. doi: 10.1093/bmb/ldr038. Epub 2011 Sep 4. PMID 21893483
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Fearon AM, Ganderton C, Scarvell JM, Smith PN, Neeman T, Nash C, Cook JL. Development and validation of a VISA tendinopathy questionnaire for greater trochanteric pain syndrome, the VISA-G. Man Ther. 2015 Dec;20(6):805-13. doi: 10.1016/j.math.2015.03.009. Epub 2015 Apr 2. PMID 25870117
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877